CLINICAL TRIAL: NCT03799224
Title: Decitabine Plus mBU/CY Preconditioning for Relapse/Refractory Acute Leukemia Patients Undergoing HSCT
Brief Title: Decitabine Plus mBU/CY Preconditioning for Relapse/Refractory Acute Leukemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Director of the Hematology Department, Peking University People's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: decitabine pre-HSCT for R/R AL
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Stem Cell Transplant Complications; Relapse Leukemia; Refractory Leukemia
Keywords: recurrent acute leukemia; refractory acute leukemia; preconditioning regimen; allogeneic stem cell transplantation
MeSH Terms: conditions — Leukemia | interventions — Decitabine

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this study would receive decitabine 200mg·m-2·d-1 on day -12 and -11 pre-HSCT. The conditioning therapy for human leukocyte antigen (HLA)-mismatched HSCT patients was modified BU/CY plus ATG. In matched sibling transplantations, patients received hydroxycarbamide (80 mg·kg-1) orally on day -10 and a lower dose of Ara-C (2 g·m-2·d-1) on day -9, but otherwise an identical regimen to the HLA-mismatched patients without ATG.BM samples from patients would be obtained to assess leukemia status after HSCT. The time points that we monitored BM samples included at time of allo-HSCT; 1 month, 2 months, 3 months, 4.5 months, 6 months, 9 months, and 12 months after allo-HSCT; and every 6 months thereafter to the defined endpoints or for at least until 5 year after transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decitabine plus mBU/CY for HLA-mismatched HSCT (Experimental): Decitabine plus mBU/CY as precondition regimen for recurrent and refractory acute leukemia at the time of HLA-mismatched HSCT
  Details:
  The conditioning therapy for human leukocyte antigen (HLA)-mismatched HSCT patients was decitabine plus modified BU/CY and ATG,consisting of decitabine 100mg·m-2·d-1 q12h on days-12 and -11,cytarabine (Ara-C 4 g·m-2·d-1) intravenously on days -10 to -9, busulfan (BU 3.2 mg·kg-1·d-1) intravenously on days -8 to -6, cyclophosphamide (CY 1.8 g·m-2·d-1), intravenously on days -5 to -4, semustine (Me-CCNU, 250 mg/m2), orally once on day -3, and ATG (2.5 mg·kg-1·d-1) intravenously on days -5 to -2
  Interventions: Drug: Decitabine; Drug: mBU/CY and ATG
- Decitabine plus mBU/CY for matched sibling transplant (Experimental): Decitabine plus mBU/CY as precondition regimen for High Risk Acute Leukemia With MRD (minimal residual disease) at the time of matched sibling transplant.
  Details:
  In matched sibling transplantations, patients received decitabine 100mg·m-2·d-1 q12h on days-12 and -11,hydroxycarbamide (80 mg/kg) orally on day -10 and a lower dose of Ara-C (2 g·m-2·d-1) on day -9, busulfan (BU 3.2 mg·kg-1·d-1) intravenously on days -8 to -6, cyclophosphamide (CY 1.8 g·m-2·d-1), intravenously on days -5 to -4, semustine (Me-CCNU, 250 mg/m2), orally once on day -3.
  Interventions: Drug: Decitabine; Drug: mBU/CY

INTERVENTIONS:
Drug: Decitabine — Decitabine 200mg.m-2.d-1 intravenously on days -12 and -11
Drug: mBU/CY and ATG — Ara-C 4 g·m-2·d-1 intravenously on days -10 to -9 Busulfan (BU 3.2 mg·kg-1·d-1) intravenously on days -8 to -6, Cyclophosphamide (CY 1.8 g·m-2·d-1) intravenously on days -5 to -4 Semustine (Me-CCNU, 250 mg·m-2) orally once on day -3 ATG (2.5 mg·kg-1·d-1) intravenously on days -5 to -2
  Arms: Decitabine plus mBU/CY for HLA-mismatched HSCT
Drug: mBU/CY — hydroxycarbamide (80 mg·kg-1) orally on day -10 Ara-C (2 g·m-2·d-1) on day -9 Busulfan (BU 3.2 mg·kg-1·d-1) intravenously on days -8 to -6, Cyclophosphamide (CY 1.8 g·m-2·d-1) intravenously on days -5 to -4 Semustine (Me-CCNU, 250 mg·m-2) orally once on day -3
  Arms: Decitabine plus mBU/CY for matched sibling transplant

SUMMARY:
Allogeneic haematopoietic stem cell transplantation (allo-HSCT) remains one of the currently available curative therapies for acute leukemia (AL). Leukemia relapse is one of the mainly causes of transplant failure. We reported previously that patients with relapse or refractory AL were at very high risk of relapse post allo-HSCT, with cumulative relapse rate of 50-80%. Decitabine has been demonstrated efficacy in the treatment of patients with recurrent or refractory leukemia and myelodysplastic syndrome. It was reported that the combination of decitabine, with busulfan and cyclophosphamide as a preparative regimen for allo-HSCT using HLA-matching donors was safe and effective. In this prospective, single-arm clinical trial, we aimed to examine the efficacy of combining decitabine with modified busulfan and cyclophosphamide (mBU/CY) as a preparative regimen for allo-HSCT in recurrent and refractory AL patients.

DETAILED DESCRIPTION:
Patients enrolled in this study would receive decitabine 200mg·m-2·d-1 on day -12 and -11 pre-HSCT. The conditioning therapy for human leukocyte antigen (HLA)-mismatched HSCT patients was modified BU/CY plus ATG (thymoglobulin; Sang Stat, France) consisting of cytarabine (Ara-C 4 g·m-2·d-1) intravenously on days -10 to -9, busulfan (BU 3.2 mg·kg-1·d-1) intravenously on days -8 to -6, cyclophosphamide (CY 1.8 g·m-2·d-1), intravenously on days -5 to -4, semustine (Me-CCNU, 250 mg·m-2), orally once on day -3, and ATG (2.5 mg·kg-1·d-1) intravenously on days -5 to -2. In matched sibling transplantations, patients received hydroxycarbamide (80 mg·kg-1) orally on day -10 and a lower dose of Ara-C (2 g·m-2·d-1) on day -9, but otherwise an identical regimen to the HLA-mismatched patients without ATG.

BM(bone marrow) samples from patients were obtained to assess leukemia status after HSCT. The time points that we monitored BM samples included at time of allo-HSCT; 1 month, 2 months, 3 months, 4.5 months, 6 months, 9 months, and 12 months after allo-HSCT; and every 6 months thereafter to the defined endpoints or for at least until 5 years after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* patients with relapsed acute leukemia
* patients with acute leukemia in the third（or more）complete remission (CR3) status

Exclusion Criteria:

* pregnancy women
* uncontrolled severe infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
1 year cumulative incidence of relapse | 1 year post allo-HSCT
  The cumulative incidence of relapse at 1 year post allo-HSCT
2 year cumulative incidence of relapse | 2 years post allo-HSCT
  The cumulative incidence of relapse at 2 years post allo-HSCT

SECONDARY OUTCOMES:
Non-relapse mortality | 1 year post allo-HSCT
  The cumulative incidence of non-relapse mortality at 1 year post allo-HSCT
1 year overall survival | 1 year post allo-HSCT
  The overall survival at 1 year post allo-HSCT
5 years overall survival | 5 years post allo-HSCT] 1 year leukemia free survival
  The overall survival at 5 years post allo-HSCT
1 year leukemia free survival | 1 year post allo-HSCT
  The leukemia free survival at 1 years post allo-HSCT
5 years leukemia free survival | 5 years post allo-HSCT
  The leukemia free survival at 5 years post allo-HSCT
engraftment | 100 days post allo-HSCT
  The total neutrophil and platelet engraftment rate
Acute graft versus host disease | 100 days post allo-HSCT
  The cumulative incidence of grade II-IV acute graft versus host disease
Chronic graft versus host disease | 1 years post allo-HSCT
  The cumulative incidence of intermediate to severe chronic graft versus host disease

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology,Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No